CLINICAL TRIAL: NCT00205270
Title: Antibody Responses to Influenza Vaccine in Pre- and Post-lung Transplant Patients
Brief Title: Influenza Vaccine in Lung Transplant Patients
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2004-0240; A561000 (Other: UW Madison); PHARM/PHARMACY/PHARMACY (Other: UW Madison)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Influenza
Keywords: Pre or post-lung transplant; Healthy
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Pre-transplant Vaccine: Cohort consists of individuals waiting for lung transplantation. Inactivated influenza vaccine will be administered intramuscularly annually.
  Interventions: Drug: Influenza vaccine
- 0-6 Months Post-transplant Vaccine: Cohort consist of individuals who have received lung transplants and received inactivated influenza vaccine 0-6 months post transplant.
  Interventions: Drug: Influenza vaccine
- 13-60 months Post-transplant Vaccine: Cohort consist of individuals who have received lung transplants and received inactivated influenza vaccine 13-60 months post transplant.
  Interventions: Drug: Influenza vaccine
- Greater than 110 months Post-transplant Vaccine: Cohort consist of individuals who have received lung transplants and received inactivated influenza vaccine greater than 110 months post transplant.
  Interventions: Drug: Influenza vaccine
- Healthy Controls: Healthy controls to measure normal immune response to the influenza vaccine
  Interventions: Drug: Influenza vaccine

INTERVENTIONS:
Drug: Influenza vaccine — influenza vaccine 0.5 ml intramuscularly each season

SUMMARY:
This 5-year study was designed to investigate how antibody and T cell responses following influenza vaccine compare among lung transplant patients, patients waiting for lung transplantation, and healthy individuals.

DETAILED DESCRIPTION:
[Note: there are 6 ClinicalTrials.gov records associated with this study, each representing a different sub-study of the population over the 5-year period, please see NCT04533061, NCT04533139, NCT04531787, NCT04530786, and NCT04531657 for related data]

Although pre-transplant immunization is routinely recommended, this recommendation is based on little data. The primary objective of this study is to compare antibody responses in lung transplant patients who receive influenza vaccine before transplant, within the first six months of transplant, between 13 and 60 months post-transplant, and 110 months or beyond transplant.

This prospective cohort study is to include immunization events performed over five years to measure H1N1, H3N2, and B antibody responses to the influenza vaccine in pre- and post-lung transplant patients. The pre-transplant patients will move to the post-transplant group as the study progressed. Similarly, participants are allowed to move to the next time-since-transplant group as time elapsed.

Serum was collected from participants prior to and two-four weeks following trivalent inactivated influenza immunization for each season.

Geometric mean titers, seroprotection (antibody titer at least 1:40), seroconversion (fourfold increase between pre and post), and mean fold increases will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care pre- or post-lung transplant at University of Wisconsin Hospital
* Healthy adult

Exclusion Criteria:

* Allergy to eggs
* Moderate to severe febrile illness
* Active treatment for acute rejection
* Received season's influenza vaccine prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults and patients receiving care pre- or post-lung transplant at University of Wisconsin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2004-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Antibody response to influenza vaccine | Each season

SECONDARY OUTCOMES:
T cell response to influenza vaccine antigens | Each season for the first two seasons

CONTACTS AND LOCATIONS:
Overall Officials: Mary S Hayney, PharmD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dopp JM, Wiegert NA, Moran JJ, Francois ML, Radford KL, Thomas H, Love RB, Hayney MS. Effect of annual influenza immunization on antibody response in lung transplant patients. Prog Transplant. 2009 Jun;19(2):153-9. doi: 10.1177/152692480901900209. PMID 19588665
- [Result] Hayney MS, Moran J, Wiegert NA, Burlingham WJ. Lung transplant patients' T cell responses to influenza vaccine viruses between seasons. Vaccine. 2008 May 19;26(21):2596-600. doi: 10.1016/j.vaccine.2008.03.012. Epub 2008 Mar 31. PMID 18420314
- [Result] Moran JJ, Rose WE, Darga AJ, Rohde KA, Hayney MS. Persistence of influenza vaccine-induced antibodies in lung transplant patients between seasons. Transpl Infect Dis. 2011 Oct;13(5):466-70. doi: 10.1111/j.1399-3062.2011.00654.x. Epub 2011 May 27. PMID 21615847
- [Result] Severson JJ, Richards KR, Moran JJ, Hayney MS. Persistence of influenza vaccine-induced antibody in lung transplant patients and healthy individuals beyond the season. Hum Vaccin Immunother. 2012 Dec 1;8(12):1850-3. doi: 10.4161/hv.21735. Epub 2012 Aug 21. PMID 22906937
- [Result] Long AJ, Worzella SL, Moran JJ, Hayney MS. Influenza vaccine antibody response and 6-month persistence in lung transplant recipients using two definitions of seroprotection. Transplantation. 2015 Apr;99(4):885-9. doi: 10.1097/TP.0000000000000391. PMID 25148380
- [Result] Miller RM, Rohde KA, Tingle MT, Moran JJ, Hayney MS. Antibody responses to influenza vaccine in pre- and post-lung transplant patients. Clin Transplant. 2016 May;30(5):606-12. doi: 10.1111/ctr.12726. Epub 2016 Mar 20. PMID 26928266